CLINICAL TRIAL: NCT06734286
Title: CogMed Intervention Targeting Working Memory in Patients with Mild Cognitive Impairment
Brief Title: Working Memory Training in Patients with Mild Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: Barrow Neurological Foundation (Other); Barrow Neurological Institute (Other)
Responsible Party: Principal Investigator, Yonas Geda, Principal Investigator, M.D., St. Joseph's Hospital and Medical Center, Phoenix
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 24-500-385-30-53
Record Dates: First submitted 2024-11-21; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-11

CONDITIONS: Mild Cognitive Impairment (MCI)
Keywords: CogMed; Mild cognitive Impairment; CogMed intervention targeting working memory; CogMed Intervention Vs Treatment as Usual; working memory training; Alzheimer's Disease
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: In this study, participant randomization into intervention and control groups will be performed using computer-generated random numbers. The goal is to successfully recruit 10 MCI patients (5 in the intervention group and 5 in the control group) who are willing to undergo blood draws for p-Tau 217 level determination. For ethical reason, at the end of trial at 3 months, the control group will also be offered the CogMed intervention.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): The Intervention Group (N = 5) Participants will be instructed to do CogMed intervention (computerized working memory activity carried out for 25 minutes daily for 5 days per week for a total of 10 weeks).
  Interventions: Other: CogMed
- Control Group (No Intervention): The Control group(N = 5) follow there Treatment as usual(TAU). For ethical reasons, at the end of trial, the control group will also be offered the CogMed intervention.

INTERVENTIONS:
Other: CogMed — CogMed which is a computerized working memory training program developed by Karolinska University.
  Other Names: Computer based training program.; CogMed Intervention.
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to test whether a special memory training program, called CogMed, can help people with early memory problems. The Investigators want to see if this training improves memory and also helps reduce stress.

The Investigators also want to see if CogMed results in changes to a blood biomarker called p-Tau 217, which possibly indicate Alzheimer's disease (AD).

DETAILED DESCRIPTION:
The goal of this study is to conduct a pilot clinical trial aimed at comparing the effects of CogMed intervention plus Treatment As Usual (TAU) versus TAU alone in patients with Mild Cognitive Impairment (MCI). Based on our preliminary data from brain health program, the primary hypothesis is that the CogMed intervention may improve the CogMed measures and possibly working memory. This may improve sense of self-efficacy and lead to a decrease in perceived stress, thereby demonstrating possible transfer of cognitive benefits to biobehavioral construct of perceived stress. Additionally, the study aims to demonstrate the feasibility of collecting p-Tau 217, a blood based Alzheimer's Disease biomarker, from MCI patients. Though no significant changes in pTau 217 are expected due to the short duration of the study, the goal is to successfully recruit 10 MCI patients (5 in the intervention group and 5 in the control group) who are willing to undergo blood draws for p-Tau 217 level determination.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female outpatients ages ≥ 50 years;
2. Meet Mayo Clinic Criteria for MCI. (Patients with mild cognitive impairment)
3. Access to the internet through computer
4. A proficiency in speaking and reading English or having a family member who is proficient in reading and speaking English and is willing to serve as a translator.
5. Vision and hearing must be sufficient to comply with study procedures.

Exclusion Criteria:

1. Mini Mental State Exam (MMSE) score less than 19 or patients diagnosed with moderate or severe dementia by a clinician.
2. In the opinion of the investigator, participation would not be in the best interest of the subject.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Working Memory as measured by the WAIS-IV Digit Span Forward/Backward | Will be assessed at baseline and again at a 3-month follow-up following the intervention period.
  The Digit Span Forward/Backward is a subset of the Wechsler Adult Intelligence Scale (WAIS) that captures attention efficiency and working memory.
Working Memory as measured by the TMT-B | Will be assessed at baseline and again at a 3-month follow-up following the intervention period.
  The Trail Making Test (TMT) is a well-established test sensitive to impairment in multiple cognitive domains.
Working Memory as measured by Category Fluency Test | Will be assessed at baseline and again at a 3-month follow-up following the intervention period.
  The Category Fluency Test (CFT) was created to assess semantic fluency. It consists of asking the individual to name as many animals as possible in 60 s. Performance on CFT can be evaluated through several components, such as the number of correct words, clusters, switching, related words, and intrusion and perseveration errors.

SECONDARY OUTCOMES:
Change in Blood biomarker | Will be assessed at baseline and again at a 3-month follow-up following the intervention period.
  We do not expect a significant change in p-Tau 217 during the short-proposed study duration, however, we projected that we will successfully recruit 10 MCI patients (Intervention group = N 5; and control group (N=5) that will be willing to undergo blood draw for determination of p-Tau 217 level.
Perceived Stress Scale (PSS) Score | Will be assessed at baseline and again at a 3-month follow-up following the intervention period.
  The Perceived Stress Scale (PSS) is used for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful. The scale also includes questions about current levels of experienced stress (Cohen et al, 1983).
Brief Resilience Scale (BRS) Score | Will be assessed at baseline and again at a 3-month follow-up following the intervention period.
  The Brief Resilience Scale (BRS) has 6 items and is a reliable means of assessing resilience as the ability to bounce back or recover from stress (Smith et al., 2008).
Pittsburgh Sleep Quality Index (PSQI) Score | Will be assessed at baseline and again at a 3-month follow-up following the intervention period.
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire designed to measure sleep quality and disturbance over past month (Buysse et al.,1989).
Physical Activity and Sedentary Behavior Questionnaire Score | Will be assessed at baseline and again at a 3-month follow-up following the intervention period.
  The Physical Activity and Sedentary Behavior Questionnaire will assess active time and time spent on exercise (PASB-Q; English Version) (Sattler et al., 2020).
Mediterranean Diet Scale(MedDiet) | Will be assessed at baseline and again at a 3-month follow-up following the intervention period.
  The MDScale includes nine components, including beneficial components (i.e., vegetables, legumes, fruits and nuts, cereal, and fish), detrimental components (i.e., meat, poultry, and high-fat dairy products), ethanol intake, and the ratio of monounsaturated to saturated fatty acids.
WHO Quality of Life Questionnaire | Will be assessed at baseline and again at a 3-month follow-up following the intervention period.
  The WHO QOL has four domains (physical health, psychological, social relationships, and environment). The four domain scores denote an individual's perception of quality of life in each particular domain (WHOQOL Group, 1998).
Memory as measured by the Comprehensive Trail Making Test (CTMT) | Will be assessed at baseline and again at a 3-month follow-up following the intervention period.
  The Comprehensive Trail Making Test (CTMT) is a measure of organized visual search, attention, set shifting and divided attention (Reynolds 2002).
Cognitive Impairment as measured by the Mini Mental State Examination (MMSE) | Will be assessed at baseline and again at a 3-month follow-up following the intervention period.
  The Mini Mental State Examination (MMSE) is used extensively in clinical and research settings to systematically measure and assess mental status. It is an 11- question measure that tests five areas of cognitive function: orientation, registration, attention, and calculation, recall, and language (Folstein et al., 1975)
Verbal Memory as Measured by the Auditory Verbal Learning Test (AVLT) | Will be assessed at baseline and again at a 3-month follow-up following the intervention period.
  The Auditory Verbal Learning Test (AVLT) evaluates verbal memory by presenting a 15- word list five times followed by attempted recall. This is followed by a second 15-word recall interference list, followed by recall of the original list (Rey A. 1964).
Comprehensive Assessment of Acceptance and Commitment Therapy Process (CompACT) | Will be assessed at baseline and again at a 3-month follow-up following the intervention period.
  The Comprehensive Assessment of Acceptance and Commitment Therapy Process (CompACT) is a 23 item questionnaire that measures ACT processes, including psychological flexibility (Francis et al., 2016).

CONTACTS AND LOCATIONS:
Overall Officials: Yonas E Geda, M.D, MSc, Principal Investigator — Barrow Neurological Institute, Alzheimer's Disease and Cognitive Disorders Division
Locations (1):
- Barrow Neurological Institute, Division of Alzheimer's Disease, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
This project will be submitted for abstracts and/or publications following data analysis. If the findings are significant a follow up study will be proposed by applying to the NIH for additional grant funding.

REFERENCES:
- [Background] Apiquian R, Diaz R, Victoria G, Ulloa RE. The Category Fluency Test components and their association with cognition and symptoms in adolescents with schizophrenia. Schizophr Res Cogn. 2023 Nov 10;35:100296. doi: 10.1016/j.scog.2023.100296. eCollection 2024 Mar. PMID 38025823
- [Background] Kortte KB, Horner MD, Windham WK. The trail making test, part B: cognitive flexibility or ability to maintain set? Appl Neuropsychol. 2002;9(2):106-9. doi: 10.1207/S15324826AN0902_5. PMID 12214820
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712
- [Background] Flak MM, Hol HR, Hernes SS, Chang L, Engvig A, Bjuland KJ, Pripp A, Madsen BO, Knapskog AB, Ulstein I, Lona T, Skranes J, Lohaugen GCC. Adaptive Computerized Working Memory Training in Patients With Mild Cognitive Impairment. A Randomized Double-Blind Active Controlled Trial. Front Psychol. 2019 Apr 12;10:807. doi: 10.3389/fpsyg.2019.00807. eCollection 2019. PMID 31031677
- [Background] Wilson, K. G., Sandoz, E. K., Kitchens, J., & Roberts, M. E. (2010). "The Valued Living Questionnaire: Defining and measuring valued action within a behavioral framework." The Psychological Record 60: 249-272
- [Background] Reynolds, C. R. (2002). Comprehensive trail-making test : examiner's manual. Austin, Tex., Pro-Ed
- [Background] Rey, A. (1964). L'examen clinique en psychologie. Paris, Presses Universitaires de France
- [Background] Francis, A. W., D. L. Dawson and N. Golijani-Moghaddam (2016). "The development and validation of the Comprehensive assessment of Acceptance and Commitment Therapy processes (CompACT)." Journal of Contextual Behavioral Science 5(3): 134-145
- [Background] Wechsler, D. (1997). Wechsler Adult Intelligence Scale-III. New York, The Psychological Corporation.
- [Background] Westwood AJ, Beiser A, Jain N, Himali JJ, DeCarli C, Auerbach SH, Pase MP, Seshadri S. Prolonged sleep duration as a marker of early neurodegeneration predicting incident dementia. Neurology. 2017 Mar 21;88(12):1172-1179. doi: 10.1212/WNL.0000000000003732. Epub 2017 Feb 22. PMID 28228567
- [Background] Smith BW, Dalen J, Wiggins K, Tooley E, Christopher P, Bernard J. The brief resilience scale: assessing the ability to bounce back. Int J Behav Med. 2008;15(3):194-200. doi: 10.1080/10705500802222972. PMID 18696313
- [Background] Simons DJ, Boot WR, Charness N, Gathercole SE, Chabris CF, Hambrick DZ, Stine-Morrow EA. Do "Brain-Training" Programs Work? Psychol Sci Public Interest. 2016 Oct;17(3):103-186. doi: 10.1177/1529100616661983. PMID 27697851
- [Background] Sattler MC, Jaunig J, Tosch C, Watson ED, Mokkink LB, Dietz P, van Poppel MNM. Current Evidence of Measurement Properties of Physical Activity Questionnaires for Older Adults: An Updated Systematic Review. Sports Med. 2020 Jul;50(7):1271-1315. doi: 10.1007/s40279-020-01268-x. PMID 32125670
- [Background] Norton MC, Clark CJ, Tschanz JT, Hartin P, Fauth EB, Gast JA, Dorsch TE, Wengreen H, Nugent C, Robinson WD, Lefevre M, McClean S, Cleland I, Schaefer SY, Aguilar S. The design and progress of a multidomain lifestyle intervention to improve brain health in middle-aged persons to reduce later Alzheimer's disease risk: The Gray Matters randomized trial. Alzheimers Dement (N Y). 2015 May 16;1(1):53-62. doi: 10.1016/j.trci.2015.05.001. eCollection 2015 Jun. PMID 29854925
- [Background] Marengoni A, Winblad B, Karp A, Fratiglioni L. Prevalence of chronic diseases and multimorbidity among the elderly population in Sweden. Am J Public Health. 2008 Jul;98(7):1198-200. doi: 10.2105/AJPH.2007.121137. Epub 2008 May 29. PMID 18511722
- [Background] Livingston G, Sommerlad A, Orgeta V, Costafreda SG, Huntley J, Ames D, Ballard C, Banerjee S, Burns A, Cohen-Mansfield J, Cooper C, Fox N, Gitlin LN, Howard R, Kales HC, Larson EB, Ritchie K, Rockwood K, Sampson EL, Samus Q, Schneider LS, Selbaek G, Teri L, Mukadam N. Dementia prevention, intervention, and care. Lancet. 2017 Dec 16;390(10113):2673-2734. doi: 10.1016/S0140-6736(17)31363-6. Epub 2017 Jul 20. No abstract available. PMID 28735855
- [Background] Krell-Roesch J, Vemuri P, Pink A, Roberts RO, Stokin GB, Mielke MM, Christianson TJ, Knopman DS, Petersen RC, Kremers WK, Geda YE. Association Between Mentally Stimulating Activities in Late Life and the Outcome of Incident Mild Cognitive Impairment, With an Analysis of the APOE epsilon4 Genotype. JAMA Neurol. 2017 Mar 1;74(3):332-338. doi: 10.1001/jamaneurol.2016.3822. PMID 28135351
- [Background] Krell-Roesch J, Syrjanen JA, Vassilaki M, Barisch-Fritz B, Trautwein S, Boes K, Woll A, Kremers WK, Machulda MM, Mielke MM, Knopman DS, Petersen RC, Geda YE. Association of non-exercise physical activity in mid- and late-life with cognitive trajectories and the impact of APOE epsilon4 genotype status: the Mayo Clinic Study of Aging. Eur J Ageing. 2019 Apr 12;16(4):491-502. doi: 10.1007/s10433-019-00513-1. eCollection 2019 Dec. PMID 31798373
- [Background] Krell-Roesch J, Pink A, Roberts RO, Stokin GB, Mielke MM, Spangehl KA, Bartley MM, Knopman DS, Christianson TJ, Petersen RC, Geda YE. Timing of Physical Activity, Apolipoprotein E epsilon4 Genotype, and Risk of Incident Mild Cognitive Impairment. J Am Geriatr Soc. 2016 Dec;64(12):2479-2486. doi: 10.1111/jgs.14402. Epub 2016 Nov 1. PMID 27801933
- [Background] Krell-Roesch J, Feder NT, Roberts RO, Mielke MM, Christianson TJ, Knopman DS, Petersen RC, Geda YE. Leisure-Time Physical Activity and the Risk of Incident Dementia: The Mayo Clinic Study of Aging. J Alzheimers Dis. 2018;63(1):149-155. doi: 10.3233/JAD-171141. PMID 29614667
- [Background] Jack CR Jr, Bennett DA, Blennow K, Carrillo MC, Dunn B, Haeberlein SB, Holtzman DM, Jagust W, Jessen F, Karlawish J, Liu E, Molinuevo JL, Montine T, Phelps C, Rankin KP, Rowe CC, Scheltens P, Siemers E, Snyder HM, Sperling R; Contributors. NIA-AA Research Framework: Toward a biological definition of Alzheimer's disease. Alzheimers Dement. 2018 Apr;14(4):535-562. doi: 10.1016/j.jalz.2018.02.018. PMID 29653606
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Hachinski V, Einhaupl K, Ganten D, Alladi S, Brayne C, Stephan BCM, Sweeney MD, Zlokovic B, Iturria-Medina Y, Iadecola C, Nishimura N, Schaffer CB, Whitehead SN, Black SE, Ostergaard L, Wardlaw J, Greenberg S, Friberg L, Norrving B, Rowe B, Joanette Y, Hacke W, Kuller L, Dichgans M, Endres M, Khachaturian ZS. Preventing dementia by preventing stroke: The Berlin Manifesto. Alzheimers Dement. 2019 Jul;15(7):961-984. doi: 10.1016/j.jalz.2019.06.001. PMID 31327392
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Brookmeyer R, Gray S, Kawas C. Projections of Alzheimer's disease in the United States and the public health impact of delaying disease onset. Am J Public Health. 1998 Sep;88(9):1337-42. doi: 10.2105/ajph.88.9.1337. PMID 9736873
- See also: World Health Organization (2017). "Global action plan on the public health response to dementia 2017-2025." — https://www.who.int/publications/i/item/global-action-plan-on-the-public-health-response-to-dementia-2017---2025